CLINICAL TRIAL: NCT00176670
Title: Is Preoperative Distraction With a Hand Held Game Boy as Effective as Midazolam in Reducing Preoperative Anxiety Levels in Children?
Brief Title: A GameBoy as a Distraction Before Surgery in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Responsible Party: Anuradha patel, MD, UMDNJ-Newark
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0120030315
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2008-06

CONDITIONS: Anxiety
Keywords: presurgical anxiety, children,
MeSH Terms: conditions — Anxiety Disorders | interventions — Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: midazolam or GameBoy or parental presence

SUMMARY:
Preoperative anxiety is characterized by subjective feelings of tension, apprehension, nervousness and worry. In children, preoperative anxiety is reported to result in postoperative negative psychological effects, including nightmares, separation anxiety, eating problems and increased fear of doctors. Anxiety in children can be expressed in many forms. Many children look scared, become agitated, breathe deeply, tremble, and stop talking or playing and start to cry. They may unexpectedly urinate or may actively attempt to escape from the medical personnel. These reactions reflect the child's fear of separation from the parents, as well as loss of control, unfamiliar routines, instruments and hospital procedures [1].

Previous studies have assessed anxiety in children during the preoperative period and the effects of premedication and parental presence during induction of anesthesia (PPIA) [2]. Midazolam has been proven to reduce preoperative anxiety in children [3]. Side effects related to oral midazolam administered to healthy children are minimal and the drug can be reversed with flumazenil but post operative recovery may be delayed in those children undergoing a short surgical procedure. It is the experience of the investigator that there are some children who have such low levels of anxiety they do not require any intervention

Distraction may be particularly helpful in children ages 6-12 as these children may not receive preoperative medication due to their curiosity about the environment. Previous studies regarding distraction therapy have focused on the parent either blowing bubbles or reading to a child [4]. Studies where the child is actively engaged in a distraction activity have not been documented.

The purpose of this investigation is to determine whether in the presence of a parent an interactive distraction intervention, i.e. Game Boy which is a hand held video game, is as effective as preoperative Midazolam in reducing preoperative anxiety. This study may help in the search for a low cost and easy to implement method of reducing anxiety for children undergoing surgery.

DETAILED DESCRIPTION:
Preoperative anxiety is characterized by subjective feelings of tension, apprehension, nervousness and worry. In children, preoperative anxiety is reported to result in postoperative negative psychological effects, including nightmares, separation anxiety, eating problems and increased fear of doctors. Anxiety in children can be expressed in many forms. Many children look scared, become agitated, breathe deeply, tremble, and stop talking or playing and start to cry. They may unexpectedly urinate or may actively attempt to escape from the medical personnel. These reactions reflect the child's fear of separation from the parents, as well as loss of control, unfamiliar routines, instruments and hospital procedures [1].

Previous studies have assessed anxiety in children during the preoperative period and the effects of premedication and parental presence during induction of anesthesia (PPIA) [2]. Midazolam has been proven to reduce preoperative anxiety in children [3]. Side effects related to oral midazolam administered to healthy children are minimal and the drug can be reversed with flumazenil but post operative recovery may be delayed in those children undergoing a short surgical procedure. It is the experience of the investigator that there are some children who have such low levels of anxiety they do not require any intervention

Distraction may be particularly helpful in children ages 6-12 as these children may not receive preoperative medication due to their curiosity about the environment. Previous studies regarding distraction therapy have focused on the parent either blowing bubbles or reading to a child [4]. Studies where the child is actively engaged in a distraction activity have not been documented.

The purpose of this investigation is to determine whether in the presence of a parent an interactive distraction intervention, i.e. Game Boy which is a hand held video game, is as effective as preoperative Midazolam in reducing preoperative anxiety. This study may help in the search for a low cost and easy to implement method of reducing anxiety for children undergoing surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ages 4 years to 16 years
2. ASA rating of I-II
3. Mask induction of general anesthesia

Exclusion Criteria:

1. Emergency Surgery
2. Children who have developmental disabilities or chronic illness
3. Children who have had repetitive surgeries.
4. Families who do not have a telephone

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 158
Dates: Start 2004-01; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Yale Preoperative Anxiety Scale

SECONDARY OUTCOMES:
10-14 days post hospitalization behavioral questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Anuradha Patel, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- New Jersey Medical School, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No